CLINICAL TRIAL: NCT00516035
Title: Phase 1 Inpatient Study of the Safety and Immunogenicity of Live Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/Chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca), a Live Attenuated Virus Vaccine Candidate for the Prevention of Avian Influenza H7N3 Infection in the Event of a Pandemic
Brief Title: Single Group Study of the Safety of and Immune Response to a Bird Flu Vaccine (H7N3) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Kawsar Talaat, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 241; WIRB Protocol Number 20071381
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Influenza; Virus Diseases
Keywords: Bird Flu
MeSH Terms: conditions — Influenza, Human; Virus Diseases; Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 0.50 ml (0.25 ml in each nostril) of Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca) administered by nasal spray at two timepoints (at study entry and between Weeks 4 and 8)
  Interventions: Biological: Live Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca)

INTERVENTIONS:
Biological: Live Influenza A Vaccine H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca) — Vaccine given by nasal spray

SUMMARY:
Over the past decade, avian influenza (AI) has become a major health concern. The development of safe and effective vaccines against avian strains infecting people is important. The purpose of this study is to determine the safety of and immune response to a new AI vaccine in healthy adults against the H7N3 strain of avian influenza.

DETAILED DESCRIPTION:
The current pandemic risk associated with avian influenza H7N3 infection is significant as an increasing number of humans are infected. H7 influenza transmission usually occurs in humans when they are exposed through direct contact to infected poultry or surfaces and objects contaminated by infected poultry feces. A pandemic occurs when a new influenza subtype emerges that infects humans, causes serious illness, and spreads easily between humans. The development of a safe and effective vaccine is necessary, should a pandemic occur. The purpose of this study is to evaluate the safety and immunogenicity of a live, attenuated AI virus vaccine, H7N3 (6-2) AA ca Recombinant (A/chicken/British Columbia/CN-6/2004 x A/Ann Arbor/6/60 ca).

This study will last approximately 90 days. Participation in this study includes two 12-day hospital stays in an isolation unit at the Johns Hopkins Bayview Medical Center. All participants will receive two doses of vaccine in nasal spray form, at study entry and sometime between 4 and 8 weeks after initial vaccination. Participants will be admitted to the isolation unit 2 days prior to each vaccination. A targeted physical exam, vital signs measurement, and a nasal wash will occur daily following each vaccination until discharge. Participants will be discharged after three consecutive nasal washes on or after Day 6 are negative. Blood and urine collection will occur at selected timepoints throughout the study. A follow-up outpatient visit will occur approximately 4 weeks following each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Available for the duration of the trial
* Willing to use acceptable forms of contraception for the duration of the study

Exclusion Criteria:

* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may affect study participation
* Previously enrolled in an H7N3 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H7N3 influenza A virus (serum hemagglutination inhibition [HI] titer greater than 1:8)
* Illegal drug use or dependency determined by urine test
* Medical, work, or family problems as a result of alcohol or illicit drug use within 12 months prior to study entry
* History of severe allergic reaction
* Allergy to oseltamivir
* Asthma or reactive airways disease within 2 years prior to study entry
* History of Guillain-Barre syndrome
* HIV infected
* Hepatitis C virus infected
* Positive for hepatitis B surface antigen (HBsAg)
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to vaccination. Participants who have used topical corticosteroids are not excluded.
* Live vaccines within 4 weeks prior to study vaccination
* Killed vaccines within 2 weeks prior to study vaccination
* Absence of spleen
* Blood products within 6 months prior to study vaccination
* Current smoker unwilling to stop smoking for the duration of the study
* Have traveled to the Southern Hemisphere, Asia, or the United Kingdom within 14 days prior to study vaccination
* Have traveled on a cruise ship within 14 days prior to study vaccination
* Work in the poultry industry
* Other investigational vaccine or drug within 30 days prior to study vaccination
* Allergy to eggs or egg products
* Purified protein derivative (PPD) positive (positive tuberculosis [TB] test)
* Have family member with immunodeficiency
* Other condition that, in the opinion of the investigator, may interfere with the study
* Pregnancy or breastfeeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety, defined as the frequency of vaccine-related reactogenicity events that occur during the acute monitoring (inpatient) phase of the study | Daily for 9 days after vaccination
Immunogenicity, determined by anti-H7N3 antibody titer | Before the first vaccination, 28 days after the first vaccination but before the second vaccination, and 28 days after the second vaccination
Quantifying the amount of vaccine virus shed by each recipient; and determining the amount of serum and nasal wash antibody induced by the vaccine | Daily for 9 days after vaccination

SECONDARY OUTCOMES:
To determine the number of vaccinees infected with the vaccine virus | Daily for 8 days after each vaccination
To determine the phenotypic stability of the vaccine virus | Throughout study
To determine whether immunogenicity is enhanced by a second dose of vaccine | At study completion
To evaluate T-cell mediated and innate immune responses against the vaccine virus | Throughout study
To develop a serum bank to evaluate future H7 influenza vaccines | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research Inpatient Unit, Mason F. Lord Building, 4940 Eastern Avenue, Baltimore, Maryland, United States

REFERENCES:
- [Background] Alexander DJ. Avian influenza viruses and human health. Dev Biol (Basel). 2006;124:77-84. PMID 16447497
- [Background] Joseph T, McAuliffe J, Lu B, Jin H, Kemble G, Subbarao K. Evaluation of replication and pathogenicity of avian influenza a H7 subtype viruses in a mouse model. J Virol. 2007 Oct;81(19):10558-66. doi: 10.1128/JVI.00970-07. Epub 2007 Jul 18. PMID 17634234
- [Background] Skowronski DM, Li Y, Tweed SA, Tam TW, Petric M, David ST, Marra F, Bastien N, Lee SW, Krajden M, Brunham RC. Protective measures and human antibody response during an avian influenza H7N3 outbreak in poultry in British Columbia, Canada. CMAJ. 2007 Jan 2;176(1):47-53. doi: 10.1503/cmaj.060204. PMID 17200390
- [Derived] Talaat KR, Karron RA, Callahan KA, Luke CJ, DiLorenzo SC, Chen GL, Lamirande EW, Jin H, Coelingh KL, Murphy BR, Kemble G, Subbarao K. A live attenuated H7N3 influenza virus vaccine is well tolerated and immunogenic in a Phase I trial in healthy adults. Vaccine. 2009 Jun 8;27(28):3744-53. doi: 10.1016/j.vaccine.2009.03.082. Epub 2009 Apr 17. PMID 19464558